CLINICAL TRIAL: NCT04182061
Title: Internet-Delivered Transdiagnostic CBT Program to Improve Access for Treatment of Anxiety and Depression in Adolescents: A Randomized Controlled Trial
Brief Title: Internet Transdiagnostic-CBT for Anxiety and Depression in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSandin
Record Dates: First submitted 2019-11-20; First posted 2019-12-02 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2022-11

CONDITIONS: Anxiety Disorder; Depressive Disorder; Emotional Disorder
Keywords: Transdiagnostic-CBT, anxiety, Depression, Internet-Delivered
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Depression | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The AMTE Protocol (Experimental): Will receive the AMTE ("Aprende a Manejar tus Emociones") Protocol; this is a modified UP-A adapted as an internet-based program of T-CBT, consisting in 10 modules delivered over 12 weeks.
  Interventions: Behavioral: The AMTE protocol
- Waiting List Control Group (No Intervention): Participants in a 12-week waiting list control condition. They will be offered the possibility of receiving the online treatment protocol after the waiting list period.

INTERVENTIONS:
Behavioral: The AMTE protocol — The AMTE program is an adaptation of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A; Ehrenreich-May et al., 2018) to be applied as an internet-based protocol. Like the UP-A, the program AMTE implements a set of core principles to address common factors underling youth anxiety and depressive symptoms. It includes the following 10 modules: (1) Understanding emotional problems and disorders, (2) Getting to know your emotions and behaviors, (3) Enjoy your positive activities, (4) Mindful emotion awareness, (5) Being flexible in your thinking, (6) Confronting physical sensations, (7) Situational emotion exposure, (8) How to regulate the emotional avoidance, (9) Respiratory relaxation training, and (10) Relapse prevention.
  Other Names: "Aprende a Manejar tus Emociones" (AMTE) Protocol
  Arms: The AMTE Protocol

SUMMARY:
This study represents the first research program to assess the efficacy of transdiagnostic cognitive behavior therapy (T-CBT) delivered via internet for anxiety and depression in adolescents. The primary aim of the study was to implement the program AMTE (Aprende a Manejar tus Emociones [Learn to Manage Your Emotions]), an internet delivered T-CBT protocol designed to target both anxiety and depression symptoms and disorders (major depression disorder, dysthymic disorder, panic disorder, agoraphobia, generalized anxiety disorder, and social anxiety disorder) in adolescents, and to establish its preliminary efficacy on anxiety and depressive symptomatology. A secondary objective is to demonstrate its potential effect regarding: (a) transdiagnostic measures associated with etiology of emotional disorders including negative affect, anxiety sensitivity, and emotional avoidance, and (b) positive factors including satisfaction with life and positive affect. It is expected that the T-CBT condition will be more effective than the waitlist (WL) control group on the primary (anxiety and depression) and secondary (transdiagnostic and positive factors) outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Having identified Spanish as the first official language spoken and having good reading comprehension in Spanish.
* Reliable internet access.
* Meeting the DSM-IV diagnosis criteria for more than one emotional disorder (separation anxiety disorder, panic disorder, agoraphobia, social anxiety disorder, generalized anxiety disorder, specific phobia, major depression disorder, and dysthymia).
* No current participating in cognitive-behavioral therapy.
* No changes in medication for 4 weeks prior to the study; no changes in medication for the next 3 months.

Exclusion Criteria:

* Presence of psychotic symptoms or severe depression.
* Being diagnosed an alcohol and/or substance dependence disorder.
* The presence of high suicidal risk.
* A medical condition which prevents the participant from carry out the psychological treatment.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change on The Revised Child Anxiety and Depression Scale-30 (RCADS-30; Sandín et al., 2010) at pre, post-intervention and 3, 6 and 12 months follow-up. | Up to 12 months.
  Symptoms of anxiety (panic disorder, social phobia, separation anxiety disorder, generalized anxiety disorder, and obsessive-compulsive disorder) and depressive disorders symptoms.
Change on The Anxiety Scale for Children and Adolescents [Escala de Ansiedad para Niños y Adolescentes] (EAN; Sandín et al., 2016) at pre, post-intervention and 3, 6 and 12 months follow-up. | Up to 12 months.
  Symptoms of anxiety.
Change on The Depression Questionnaire for Children and Adolescents [Cuestionario de Depresión para Niños y Adolescentes] (CDN; Sandín et al., 2016) at pre, post-intervention and 3, 6 and 12 months follow-up. | Up to 12 months.
  Symptoms of depression.

SECONDARY OUTCOMES:
Change on The Children Positive and Negative Affect Schedule [Escalas PANAS para niños y adolescentes] (PANASN; Sandín, 2003) at pre, post-intervention and 3, 6 and 12 months follow-up. | Up to 12 months.
  Positive and negative (neuroticism) affectivity.
Change on The Childhood Anxiety Sensitivity Index (CASI) (Silverman et al.,1991) at pre, post-intervention and 3, 6 and 12 months follow-up. | Up to 12 months.
  Anxiety sensitivity.
Change on The Emotional Avoidance Strategy Inventory for Adolescents (EASI-A; Kennedy & Ehrenreich-May, 2016) at pre, post-intervention and 3, 6 and 12 months follow-up. | Up to 12 months.
  Emotional avoidance.
Change on The Satisfaction with Life Scale for Children (SWLS-C; Sandín et al., 2015) at pre, post-intervention and 3, 6 and 12 months follow-up. | Up to 12 months.
  Life satisfaction.
Change on The Pen State Worry Questionnaire (PSWQ; Meyer, Miller, Metzger, & Borkovec, 1990) adapted for children and adolescents (PSWQ-11) at pre, post-intervention and 3, 6 and 12 months follow-up. | Up to 12 months.
  Symptoms of pathological worry.
Change on The Social Anxiety Scale for Children-Revised (SASC-R; La Greca & Stone, 1993) at pre, post-intervention and 3, 6 and 12 months follow-up. | Up to 12 months.
  Symptoms of social anxiety.
Change on The Self-Reported Panic Disorder Severity Scale (PDSS-SR; Houck, Spiegel, Shear, & Rucci, 2002) at pre, post-intervention and 3, 6 and 12 months follow-up. | Up to 12 months.
  Symptoms of panic disorder severity.

CONTACTS AND LOCATIONS:
Overall Officials: Bonifacio Sandín, Ph.D., Principal Investigator — Universidad Nacional de Educación a Distancia, Madrid, Spain; Paloma Chorot, Ph.D., Principal Investigator — Universidad Nacional de Educación a Distancia, Madrid, Spain; Rosa M. Valiente, Ph.D., Study Chair — Universidad Nacional de Educación a Distancia, Madrid, Spain
Locations (1):
- Bonifacio Sandín, Madrid, Spain